CLINICAL TRIAL: NCT02636764
Title: Influence of Using Physical Therapy Resources for Knee Osteoarthritis
Acronym: osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Phd, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 51391715.1.0000.5511
Record Dates: First submitted 2015-12-10; First posted 2015-12-22 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Osteoarthritis; Physical Therapy Modalities
MeSH Terms: conditions — Osteoarthritis | interventions — Exercise; Electric Stimulation Therapy; Low-Level Light Therapy; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- exercise group (Active Comparator): An exercise protocol drawn up with the objective will be held to strengthen the musculature: flexor and extensor of the knee; extension, abduction, hip side rotator, using the weight and the elastic band.
  Interventions: Other: exercise
- exercise group + Ultrasound therapy (Placebo Comparator): Apart from intervening in the exercise group, an ultrasound device is used .
  Interventions: Other: exercise; Device: Ultrasound therapy
- exercise group + interferential current (Experimental): Besides the intervention of the exercise group after the exercises will be applied to interferential current through the device. Will be positioned 4 electrodes (8x5 cm), two upper and two lower (forming a square) around the center of the knee.
  Interventions: Other: exercise; Device: interferential current
- exercise group + short-wave diathermy (Experimental): Besides the intervention of the exercise group after the exercises will be applied diathermies short wave in continuous mode. For that will be used apparatus, 27.12 megahertz, by means of vulcanized rubber electrodes (12x17 cm) with gentle warming for 30 minutes.
  Interventions: Other: exercise; Device: short-wave diathermy
- exercise group + Low level laser therapy (Experimental): Apart from intervening in the exercise group, will be applied to Low level laser therapy, through the laser unit, Class 3b, gallium-aluminum-arsenide, continuous mode, wavelength: 830 nanometer, power: 30 watts.
  Interventions: Other: exercise; Device: Low level laser therapy

INTERVENTIONS:
Other: exercise — exercises designed with the objective of strengthening the musculature: flexor and extensor of the knee; extensor, abductor, lateral rotator of the hip.
Device: interferential current — The basic principle of Interferential Therapy (IFT) is to utilise the significant physiological effects of low frequency (<250pps) electrical stimulation of nerves without the associated painful and somewhat unpleasant side effects sometimes associated with low frequency stimulation
  Arms: exercise group + interferential current
Device: short-wave diathermy — Is a modality that produces deep heating via conversion of electromagnetic energy to thermal energy
  Arms: exercise group + short-wave diathermy
Device: Low level laser therapy — Laser treatment in which the energy output is low enough so that the temperature of the treated tissue does not rise above 98.6°F (36.5° C) or normal body temperature.
  Arms: exercise group + Low level laser therapy
Device: Ultrasound therapy — Ultrasound (US) is a form of mechanical energy, not electrical energy and therefore strictly speaking, not really electrotherapy at all but does fall into the Electro Physical Agents grouping.
  Arms: exercise group + Ultrasound therapy

SUMMARY:
Osteoarthritis is a chronic, multifactorial characterization, which changes in bone alignment, cartilage and structures that provide joint stability appear to be strongly correlated with the origin of this disease.This project will aim to verify the effectiveness of interferential current, short wave and low level laser therapy on an exercise program for mobility and pain in knee osteoarthritis. Blind randomized, placebo controlled. Five groups: exercise group, exercise group + Ultrasound therapy, exercise group + interferential current, exercise group + short-wave diathermy, exercise group + Low level laser therapy. Before and after the trial protocol by the following instruments: Western Ontario and McMaster Universities osteoarthritis index (WOMAC), numerical scale of pain assessment (END), Visual Analogue Scale Fatigue (VAS-F), issue F2.2 Instrument assessment of quality of life of the World Health Organization (WHOQOL-100) test sitting and standing + numerical rating pain scale, algometry. This project hypothesizes that the inclusion of photothermal and electrical agents in an exercise program will provide an improvement in pain, mobility and knee function in individuals diagnosed with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* knee pain to at least six months and minimum of 4 points in pain scale
* Diagnosed with osteoarthritis in unilateral knee according to the criteria established by the American College of Rheumatology and confirmed by radiographic examination for identification Kellgren-Lawrence grade 2 or 3 (Kellgren & Lawrence, 1957).

Exclusion Criteria:

* Any type of physical therapy
* therapy with intra-articular corticosteroids or therapeutic chondroprotective drugs last year, before the start of the study.
* history of trauma on his knees, cognitive disorder or psychological disorder,
* neurological (sensory or motor)
* cancer
* diabetes,
* or any state of adverse acute health osteoarthritis signs of hip
* cardiopulmonary disease that prevents the conducting exercises
* require auxiliary device for performing gait.
* Yet who undertake physical activity in the last two months. Physical activity is defined as strength training and / or more than 20 minutes of aerobic activity twice a week.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12; Primary Completion 2017-09 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
pain | Change from Baseline in The Western Ontario and McMaster Universities Arthritis Index at 8 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation Knee Osteoarthritis.
stiffness | Change from Baseline in The Western Ontario and McMaster Universities Arthritis Index at 8 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation Knee Osteoarthritis.
physical functional | Change from Baseline in The Western Ontario and McMaster Universities Arthritis Index at 8 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation Knee Osteoarthritis.

SECONDARY OUTCOMES:
intensity of pain | Change from Baseline in The Numerical rating pain scale at 8 weeks
  The Numerical rating pain scale, a simple, easily administered scale evaluates the perceived intensity of pain, using an 11-point scale from 0, representing 'no pain', to 10, which is the 'worst possible pain'.
Self-perceived fatigue | Change from Baseline in the self-perceived fatigue at 8 weeks
  a visual analog scale (VAS-F).
Functional capacity for sitting and standing | Change from Baseline in The Functional capacity for sitting and standing at 8 weeks
  sitting-rising test
level of pressure pain | Change from Baseline in ThePressure Pain Threshold at 8 weeks
  Pressure Pain Threshold in the knee with algometer dynamometer.
Self-perceived fatigue | Change from Baseline in The question of F2.2 instrument for assessing quality of life World Health Organization (WHOQOL-100) at 8 weeks
  The question of F2.2 instrument for assessing quality of life World Health Organization (WHOQOL-100).

CONTACTS AND LOCATIONS:
Overall Officials: Cid André Fidelis de Paula Gomes, Phd, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Paula Gomes CAF, Politti F, de Souza Bacelar Pereira C, da Silva ACB, Dibai-Filho AV, de Oliveira AR, Biasotto-Gonzalez DA. Exercise program combined with electrophysical modalities in subjects with knee osteoarthritis: a randomised, placebo-controlled clinical trial. BMC Musculoskelet Disord. 2020 Apr 20;21(1):258. doi: 10.1186/s12891-020-03293-3. PMID 32312265
- See also: Related Info — http://www.uninove.br